CLINICAL TRIAL: NCT06778876
Title: Effect of Lavender on Sleep Quality and Insomnia Severity in Patients With Psychophysiological Insomnia
Brief Title: Effect of Lavender on Sleep Quality and Insomnia Severity in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, bülent devrim akçay, University of Health Sciences, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SBU-RSH-BDA-01
Record Dates: First submitted 2025-01-12; First posted 2025-01-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Insomnia, Psychophysiological
Keywords: insomnia; sleep quality; Sleepiness; Lavender
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleepiness | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two groups with a control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will not be informed about group assignments and will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lavender sachet group (Active Comparator): The normal procedure applied in the sleep clinic (keeping a sleep diary, sleep hygiene education) will be followed and participants will be asked to sleep with lavender sachets inside their pillows for two weeks.
  Interventions: Other: lavender sachet group
- Control group (Sham Comparator): Participants will follow the normal procedure applied (keeping a sleep diary, sleep hygiene training) in the sleep clinic and no additional intervention will be performed.
  Interventions: Other: control group

INTERVENTIONS:
Other: lavender sachet group — The normal procedure applied in the sleep clinic (keeping a sleep diary, sleep hygiene education) will be followed and participants will be asked to sleep with lavender sachets inside their pillows for two weeks.
  Arms: lavender sachet group
Other: control group — Participants will follow the normal procedure applied (keeping a sleep diary, sleep hygiene training) in the sleep clinic and no additional intervention will be performed.
  Arms: Control group

SUMMARY:
Today, psychophysiological insomnia is the most common persistent insomnia. Lavender essential oil is frequently used in the literature as an aromatherapy method to improve sleep quality. Studies have found that lavender improves sleep quality. They also emphasized that more studies are needed in this area. When the relevant literature is reviewed, no studies examining the effects of lavender oil on patients with psychophysiological insomnia were found. In this context, the aim of the study was to evaluate the effect of lavender on sleep quality and insomnia severity in patients with psychophysiological insomnia.

DETAILED DESCRIPTION:
Today, psychophysiological insomnia is the most common persistent insomnia. The patient's inability to sleep occurs as a result of repetitive negative thoughts such as the thought that he will have difficulty sleeping before going to bed and/or past experiences involving the bedroom or the night. More effort to sleep causes more wakefulness and more difficulty falling asleep.

Numerous studies have shown that insomnia seriously affects health and quality of life and can cause various problems including memory problems, depression, irritability, cardiovascular and cerebrovascular diseases, etc. Therefore, looking for effective ways to improve sleep quality is important for individual and social health. Today, drug therapy, psychotherapy, physiotherapy and cognitive-behavioral therapy are widely used treatments for insomnia. Recently, more and more studies have found that aromatherapy is one of the non-drug treatments to improve sleep quality. Lavender essential oil appears in the literature as an aromatherapy method frequently used to improve sleep quality.

Studies have found that lavender improves sleep quality. They also emphasized that more studies are needed in this area. When the relevant literature was examined, no studies were found examining the effects of lavender oil on patients with psychophysiological insomnia. In this context, the aim of the study was to evaluate the effect of lavender on sleep quality and insomnia severity in patients with psychophysiological insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Being over 65 years old
* Being diagnosed with psychophysiological insomnia,
* Knowing Turkish at a level that will allow you to read and understand the survey questions,
* Accepting to participate in the study

Exclusion Criteria:

* Having a serious physical or cognitive disability that would prevent him/her from answering the survey,
* Being under the age of 18,
* Not accepting to participate in the study,
* Being allergic to lavender,
* Having a chronic additional disease related to the respiratory system,
* Having a psychiatric or neurological additional disease,
* Using medication(s) that may affect sleep,
* Experiencing a physical activity limitation that causes bedriddenness,
* Having or contracting a disease that will affect the ability to smell.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index | two weeks
  PSQI is a 19-item scale, assessed by self-report (19 items) and spouse/roommate responses (5 items). The scale includes components such as sleep quality, duration, and disturbance, and the total score ranges from 0 to 21; a score greater than 5 indicates poor sleep quality.

SECONDARY OUTCOMES:
The Insomnia Severity Index | two weeks
  ISS is a 7-item self-report scale. The total score obtained from this scale varies between 0 and 28, and a score of 15 and above indicates clinical insomnia.
The Epworth Sleepiness Scale | two weeks
  ESS is a four-point Likert-type scale consisting of 8 items. The score range of this scale is 0 to 24, and a score of 10 and above indicates excessive daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent D. Akçay, Assoc. Prof., Principal Investigator — Saglik Bilimleri Universitesi; Mehmet Koçer, MD, Principal Investigator — Gulhane Training and Research Hospital; Duygu Akçay, Asst.Prof, Principal Investigator — Ufuk University
Locations (1):
- University of Health Sciences, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No